CLINICAL TRIAL: NCT05704049
Title: A Randomized, Phase 2, Open Label Study Evaluating Subcutaneous Administration of Isatuximab in Combination With Carfilzomib and Dexamethasone in Adult Participants With Relapsed and/or Refractory Multiple Myeloma (RRMM)
Brief Title: A Study to Investigate Subcutaneous Isatuximab in Combination With Carfilzomib and Dexamethasone in Adult Participants With Relapsed and/or Refractory Multiple Myeloma
Acronym: IZALCO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT17453; U1111-1280-5090 (Registry Identifier: ICTRP); 2023-508870-27 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; carfilzomib; Dexamethasone; montelukast; Acetaminophen; Diphenhydramine; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Cohort 1: manual administration (Experimental): Isatuximab will be administered manually for 8 minutes on Day 1 of Cycle 1 followed by 6 minutes from Day 8 of Cycle 1 and thereafter, in combination with carfilzomib and dexamethasone. Participants may receive other treatments as rescue medication or background medication.
  Interventions: Drug: Isatuximab; Drug: Carfilzomib; Drug: Dexamethasone; Drug: Dexamethasone IV; Drug: Montelukast; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Methylprednisolone
- Part 1 Cohort 2: manual administration (Experimental): Isatuximab will be administered manually for 6 minutes on Day 1 of Cycle 1 and thereafter, in combination with carfilzomib and dexamethasone. Participants may receive other treatments as rescue medication or background medication.
  Interventions: Drug: Isatuximab; Drug: Carfilzomib; Drug: Dexamethasone; Drug: Dexamethasone IV; Drug: Montelukast; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Methylprednisolone
- Part 2 Cohort 3 Randomized Cohort: OBDS to manual (Experimental): Isatuximab will be administered in combination with carfilzomib and dexamethasone. Isatuximab will be administered via OBDS from Cycle 1 to 3. For Cycle 4 to 6, the method of administration will be switched for each participant from OBDS to manual administration. From Cycle 7 and onwards, participants can choose manual or OBDS. Participants may receive other treatments as rescue medication or background medication.
  Interventions: Drug: Isatuximab; Drug: Carfilzomib; Drug: Dexamethasone; Drug: Dexamethasone IV; Drug: Montelukast; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Methylprednisolone
- Part 2 Cohort 3 Randomized Cohort: Manual to OBDS (Experimental): Isatuximab will be administered in combination with carfilzomib and dexamethasone. Isatuximab will be administered manually from Cycle 1 to 3. For Cycle 4 to 6, the method of administration will be switched for each participant from manual to OBDS administration. From Cycle 7 and onwards, participants can choose manual or OBDS. Participants may receive other treatments as rescue medication or background medication.
  Interventions: Drug: Isatuximab; Drug: Carfilzomib; Drug: Dexamethasone; Drug: Dexamethasone IV; Drug: Montelukast; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Methylprednisolone
- Part 3 Cohort 4 Randomized Cohort: OBDS to manual (Experimental): Isatuximab will be administered in combination with carfilzomib and dexamethasone. Isatuximab will be administered via OBDS from Cycle 1 to 3. For Cycle 4 to 6, the method of administration will be switched for each participant from OBDS to manual administration. From Cycle 7 and onwards, participants can choose manual or OBDS. Participants may receive other treatments as rescue medication or background medication.
  Interventions: Drug: Isatuximab; Drug: Carfilzomib; Drug: Dexamethasone; Drug: Dexamethasone IV; Drug: Montelukast; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Methylprednisolone
- Part 3 Cohort 4: Randomized Cohort: manual to OBDS (Experimental): Isatuximab will be administered in combination with carfilzomib and dexamethasone. Isatuximab will be administered manually from Cycle 1 to 3. For Cycle 4 to 6, the method of administration will be switched for each participant from manual to OBDS administration. From Cycle 7 and onwards, participants can choose manual or OBDS. Participants may receive other treatments as rescue medication or background medication.
  Interventions: Drug: Isatuximab; Drug: Carfilzomib; Drug: Dexamethasone; Drug: Dexamethasone IV; Drug: Montelukast; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Methylprednisolone
- Part 3 Cohort 5 Randomized Cohort: OBDS to manual administration in Chinese participants (Experimental): Isatuximab will be administered in combination with carfilzomib and dexamethasone. Isatuximab will be administered via OBDS from Cycle 1 to 3. For Cycle 4 to 6, the method of administration will be switched for each participant from OBDS to manual administration. From Cycle 7 and onwards, participants can choose manual or OBDS. Participants may receive other treatments as rescue medication or background medication.
  Interventions: Drug: Isatuximab; Drug: Carfilzomib; Drug: Dexamethasone; Drug: Dexamethasone IV; Drug: Montelukast; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Methylprednisolone
- Part 3 Cohort 5 Randomized Cohort: manual to OBDS administration in Chinese participants (Experimental): Isatuximab will be administered in combination with carfilzomib and dexamethasone. Isatuximab will be administered manually from Cycle 1 to 3. For Cycle 4 to 6, the method of administration will be switched for each participant from manual to OBDS administration. From Cycle 7 and onwards, participants can choose manual or OBDS. Participants may receive other treatments as rescue medication or background medication.
  Interventions: Drug: Isatuximab; Drug: Carfilzomib; Drug: Dexamethasone; Drug: Dexamethasone IV; Drug: Montelukast; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Isatuximab — Investigational medicinal product; Pharmaceutical form: Solution for Subcutaneous administration; Route of administration: Subcutaneous
Drug: Carfilzomib — Investigational medicinal product; Pharmaceutical form: Powder for solution for infusion; Route of administration: Intravenous
  Other Names: Kyprolis
Drug: Dexamethasone — Investigational medicinal product/background treatment; ATC code: H02AB02; Pharmaceutical form: Tablet; Route of administration: Oral
Drug: Dexamethasone IV — Investigational medicinal product/background treatment; ATC code: H02AB02; Pharmaceutical form: Powder for solution for infusion; Route of administration: Intravenous
Drug: Montelukast — Background Treatment; ATC code: R03DC03; Pharmaceutical form: As per local commercial product; Route of administration: Oral
Drug: Acetaminophen — Background Treatment; ATC code: N02BE01; Pharmaceutical form: As per local commercial product; Route of administration: Oral or intravenous (IV)
Drug: Diphenhydramine — Background Treatment; ATC code: R06AA02; Pharmaceutical form: As per local commercial product; Route of administration: Oral or IV
Drug: Methylprednisolone — Background Treatment/Rescue medication; ATC code: H02AB04; Pharmaceutical form: As per local commercial product; Route of administration: IV

SUMMARY:
The main purpose of this study is to measure the efficacy (Myeloma response) of subcutaneous (SC) isatuximab treatment in combination with carfilzomib and dexamethasone in adult participants with RRMM having received 1 to 3 prior lines of therapy, and to characterize the PK of isatuximab in combination with carfilzomib and dexamethasone after manual and On Body Delivery System (OBDS) administration. After confirmation of the feasibility of SC isatuximab by manual administration, patient will be randomized to 1 of the 2 delivery methods of SC isatuximab.

DETAILED DESCRIPTION:
The duration of the study for a participant will include a period for screening of up to 28 days. A cycle duration is 28 days. Participants will be allowed to continue therapy until disease progression, unacceptable adverse events (AEs), participant request to discontinue treatment, or any other reason, as well as the study treatment is commercially available and reimbursed in the participant's country, or is available from another source, whichever is first. The overall study duration will be of approximately 45 months.

ELIGIBILITY:
Inclusion Criteria:

Participants must have a documented diagnosis of multiple myeloma (MM)

* Participants with measurable disease defined as at least one of the following:

  * Serum M-protein ≥0.5 g/dL measured using serum protein immunoelectrophoresis and/or
  * Urine M-protein ≥200 mg/24 hours measured using urine protein immunoelectrophoresis and/or
  * Serum free light chain (FLC) assay: Involved FLC assay ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65).
* Participant with relapsed and/or refractory MM with at least 1 prior line of therapy and no more than 3 prior lines of therapy.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and either is not a female of childbearing potential (FCBP) or agrees to practice complete abstinence or use approved contraception methods.
* Male participants agree to practice true abstinence or agree to use approved contraception methods while receiving study treatment, during dose interruptions and at least 5 months following study treatment discontinuation, even if has undergone a successful vasectomy.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Primary refractory MM defined as participants who have never achieved at least a minimal response (MR) with any treatment during the disease course
* Participants with prior anti-CD38 treatment if: a) administered <9 months before first isatuximab administration or randomization as applicable or, b) Intolerant to the anti-CD38 previously received
* Prior treatment with carfilzomib
* Known history of allergy to captisol (a cyclodextrin derivative used to solubilize carfilzomib), prior hypersensitivity to sucrose, histidine (as base and hydrochloride salt), polysorbate 80, or any of the components (active substance or excipient) of study treatment that are not amenable to premedication with steroids, or intolerance to arginine and Poloxamer 188 that would prohibit further treatment with these agents
* Uncontrolled or active infection with hepatitis A, B, and C virus; known acquired immunodeficiency syndrome (AIDS)-related illness; active primary amyloid light chain (AL) amyloidosis
* Any severe acute or chronic medical condition which could impair the ability of the participant to participate in the study or interfere with interpretation of study results (eg, systemic infection unless specific anti-infective therapy is employed) or participant unable to comply with the study procedures.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2028-05-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) - Cohorts 1 to 3 | 6 months after the Last Participant In (LPI) i.e., approximately 16 months
  ORR defined as the proportion of participants with stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR) according to the 2016 International Myeloma Working Group (IMWG) criteria assessed by Independent Review Committee (IRC).
Maximum observed concentration (Cmax) over Cycle 1- Cohorts 4 to 5 | Cycle 1 (28 days)
Cumulative area under the curve over the first 4 weeks (AUC4weeks) of isatuximab treatment- Cohorts 4 to 5 | Cycle 1 (28 days)

SECONDARY OUTCOMES:
Proportion of participants preferring OBDS over manual administration of isatuximab SC at Day 15 of Cycle 6 | 6 months from LPI i.e., approximately 16 months
  Patient preference for method of administration defined as the proportion of participants preferring OBDS over manual administration of isatuximab SC at Day 15 of Cycle 6 using the patient experience and satisfaction questionnaire version 2 (PESQ v2).
Incidence rate of infusion reactions (IRs) | From the signing of the informed consent to 30 days following the last administration of any study treatment i.e., up to approximately 45 months
Number of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and changes in laboratory parameters | From the signing of the informed consent to 30 days following the last administration of any study treatment i.e., up to approximately 45 months
Incidence rate of injection site reactions (ISRs) | 18 months after LPI i.e., approximately 28 months
PK concentration: trough plasma concentration (Ctrough) | Cycle 2 Day 1 and Cycle 6 Day 1 (1 Cycle = 28 days)
  Blood samples will be collected for measurement of isatuximab concentrations.
Overall response rate (ORR) | 6 months after the Last Participant In (LPI) i.e., approximately 16 months
  Proportion of participants with sCR, CR, VGPR, and PR according to the 2016 IMWG criteria assessed by investigator.
Duration of response (DOR) | 6 months after the Last Participant In (LPI) i.e., approximately 16 months
  DOR defined as time from date of first IRC-determined response for participants achieving PR or better to first documentation of progressive disease (PD) determined by IRC or death, whichever occurred first, for Cohorts 1 to 3. For Cohorts 4-5, the time from date of first investigator determined response for participants achieving PR or better to first documentation of progressive disease (PD) determined by investigator or death, whichever occurred first.
Time to first response (TT1R) | 6 months after the Last Participant In (LPI) i.e., approximately 16 months
  TT1R defined as time from first investigational medicinal product (IMP) administration or randomization to first IRC determined response (PR or better) that is subsequently confirmed, for Cohorts 1 to 3. For cohorts 4-5, the time from first IMP administration or randomization to first investigator determined response (PR or better) that is subsequently confirmed.
Time to best response (TTBR) | 6 months after the Last Participant In (LPI) i.e., approximately 16 months
  TTBR defined as time from first IMP administration or randomization to first occurrence of IRC determined best response (PR or better) that is subsequently confirmed, for Cohorts 1 to 3. For cohorts 4-5, the time from first IMP administration or randomization to first occurrence of investigator determined best response (PR or better) that is subsequently confirmed.
Progression free survival (PFS) | 18 months after LPI i.e., approximately 28 months
  PFS defined as time from the date of first IMP administration or randomization to the date of first documentation of PD as determined by IRC for Cohorts 1 to 3 and by Investigator for all cohorts, or the date of death from any cause, whichever comes first.
Overall survival (OS) | 18 months after LPI i.e., approximately 28 months
  OS defined as time from the date of first IMP administration or randomization to death from any cause.
Incidence of participants with anti-drug antibodies (ADA) against isatuximab | From Cycle 1 Day 1 to follow-up (90 days from last administration) i.e., approximately 13 months (1 Cycle = 28 days)
Patient Expectations Questionnaire at Baseline (PEQ-BL v2) with isatuximab administered subcutaneously | Baseline
  PEQ-BL v2 is a participant assessed questionnaire. It will be completed at baseline prior to study treatment administration or other study related procedures. This questionnaire has been designed to assess the expectations of the participants regarding both the treatment (side effects, worth taking) and the administration method (confidence, comfortability, pain, side effects, potential time-savings), as well as to understand previous treatment experience from the participant (experience with injection methods for oncology medication).
Patient experience and satisfaction questionnaires (PESQ v2) with isatuximab administered subcutaneously | 18 months after LPI i.e., approximately 28 months
  PESQ v2 is a participant assessed questionnaire. It has been designed to follow up on participant experience and satisfaction regarding the treatment (side effects, worth taking and overall satisfaction) and the administration method (confidence, comfortability, pain, side effects, potential time-savings and overall satisfaction). The PESQ v2 includes items to assess preference on subcutaneous injection method. This questionnaire has been developed using industry standard for instrument development and has been debriefed and adapted based on qualitative interviews with oncology patients. The more general treatment expectations instrument (v1) was further adapted and debriefed with patients to assess manual and OBDS subcutaneous delivery (v2). The PESQ v2 contains a total of 9 items. There are 6 items that are administered for the duration of treatment, and 3 preference items administered only after patient experience of both manual and OBDS.
Health state utility assessed using Health Resource Utilization and Productivity Questionnaire (HRUPQ) | 18 months after LPI i.e., approximately 28 months
  Medical resource utilization and participant productivity will be collected from participants through a specific questionnaire developed by Sanofi for cohorts 1,2, 3, and 5. The data collected include number, nature (emergency or routine) and duration of hospitalizations, emergency room visits and outpatient medical encounters and employment history.
Health Related Quality of Life (HRQL) | 18 months after LPI i.e., approximately 28 months
  HRQL is assessed for cohorts 1, 2, and 3 using the European Organization for Research and Treatment of Cancer (EORTC) myeloma module with 20 items (QLQ-MY20) and EORTC quality of life questionnaire with 30 questions (QLQ-C30); a total of 50 items. The EORTC QLQ-C30 provides a comprehensive assessment of the principal HRQL dimensions identified as relevant by cancer patients. The EORTC QLQ-MY20 is to be used in conjunction with the EORTC QLQ-C30 to assess symptoms and side effects due to the treatment or the disease which impact HRQL in participants with MM.
European Quality of Life Group questionnaire with 5 dimensions and 5 levels per dimension (EQ-5D-5L) | 18 months after LPI i.e., approximately 28 months
  Health status is assessed for cohorts 1, 2, and 3, using the EQ-5D-5L, a standardized measure of health status that provides a simple, generic measure of health utility, and consists of 2 sections: descriptive and VAS. The descriptive system consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The VAS records the respondent's self-rated health on a 20 cm vertical VAS with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. This information can be used as a quantitative measure of health as judged by the individual respondents.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (23):
- Australia (2):
  - Investigational Site Number : 0360002, Wollongong, New South Wales
  - Investigational Site Number : 0360001, Melbourne, Victoria
- Brazil (3):
  - Hospital Mae de Deus Site Number : 0760002, Porto Alegre, Rio Grande do Sul
  - Clinica São Germano- Site Number : 0760003, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo- Site Number : 0760001, São Paulo
- China (7):
  - Investigational Site Number : 1560006, Changsha
  - Investigational Site Number : 1560002, Guangzhou
  - Investigational Site Number : 1560005, Nanchang
  - Investigational Site Number : 1560004, Shenyang
  - Investigational Site Number : 1560001, Tianjin
  - Investigational Site Number : 1560007, Tianjin
  - Investigational Site Number : 1560003, Wuhan
- Czechia (4):
  - Investigational Site Number : 2030002, Brno
  - Investigational Site Number : 2030004, Olomouc
  - Investigational Site Number : 2030003, Ostrava
  - Investigational Site Number : 2030001, Prague
- Greece (2):
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000002, Athens
- Japan (2):
  - Investigational Site Number : 3920001, Kashiwa, Chiba
  - Investigational Site Number : 3920002, Okayama
- Portugal (3):
  - Investigational Site Number : 6200001, Braga
  - Investigational Site Number : 6200004, Lisbon
  - Investigational Site Number : 6200005, Lisbon

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Parmar G, Capra M, Seguro F, Hungria V, Dimopoulos MA, Delimpasi S, Minarik J, Spicka I, Pour L, Marques H, Esteves G, Sunami K, Yuda J, Hajek R, Mihalyova J, Soufflet C, Yu D, Benlhassan K, Koch V, Comerford E, Cordero P, Suzan F, Quach H. Efficacy and safety of isatuximab subcutaneous plus carfilzomib and dexamethasone in patients with relapsed/refractory multiple myeloma: results of the Phase 2 study IZALCO. Blood Cancer J. 2025 Dec 27;16(1):16. doi: 10.1038/s41408-025-01436-0. PMID 41455697
- See also: ACT17453 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25214&tenant=MT_SNY_9011